CLINICAL TRIAL: NCT03772613
Title: Optimal Target of Activated Clotting Time During Percutaneous Coronary Intervention and Outcomes: The Randomized OPTIMAL-ACT Trial
Brief Title: The Randomized OPTIMAL-ACT Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shahyar M. Gharacholou, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-005209
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Anticoagulant-induced Bleeding; Coronary Syndrome
Keywords: activated clotting time; outcomes; bleeding
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina, Unstable; Hemorrhage | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low ACT Target (Active Comparator): ACT target range of 225 to 275 seconds is achieved prior to PCI if no planned glycoprotein IIb/IIIa inhibitor used
  Interventions: Drug: Unfractionated heparin
- Medium ACT Target (Active Comparator): ACT target range of 275 to 325 seconds is achieved prior to PCI if no planned glycoprotein IIb/IIIa inhibitor used
  Interventions: Drug: Unfractionated heparin
- High ACT Target (Active Comparator): ACT target range of 325 to 375 seconds is achieved prior to PCI if no planned glycoprotein IIb/IIIa inhibitor used
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Unfractionated heparin — Administration of unfractionated heparin will be assessed using the activated clotting time

SUMMARY:
The purpose of this study is to find the ideal range of the activated clotting time (ACT) during percutaneous coronary intervention (PCI) that is associated with lowering the rate of undesirable medical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Referred for coronary angiography with possible coronary revascularization or adjunctive invasive diagnostic testing (IVUS/OCT, FFR, or iFR)

Exclusion Criteria:

* Receipt of LMWH at treatment dose (not DVT prophylaxis dose) within 6 hours of coronary angiography
* Prior GP IIb/IIIa use within the previous 72 hours
* Use of warfarin (vitamin K antagonist) or direct oral anticoagulant
* Patients on LMWH bridging strategy
* PCI within prior 30 days
* Planned use of bivalirudin as the procedural anticoagulant
* Rotational atherectomy
* Excimer laser coronary angioplasty
* Chronic total occlusions
* Patients with active bleeding disorders or bleeding diathesis
* Patients with ST-segment elevation myocardial infarction
* Patient with clinical evidence of cardiogenic shock (defined as SBP<90 mmHg for ≥30 min OR support to maintain SBP ≥90 mmHg AND evidence of end-organ hypoperfusion (urine output <30 mL/h or cool extremities)
* Chronic kidney disease stage 4/5 (GFR 30 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahyar M Gharacholou, MD, MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target
Started | 61 | 61 | 58
Completed | 61 | 60 | 57
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target | Total
Number analyzed (Participants) | 61 | 61 | 58 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 68 (10) | 67 (10) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 14 | 51
  Male | 42 | 43 | 44 | 129
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 61 | 61 | 58 | 180

OUTCOME MEASURES:

1. Primary Outcome: Bleeding
Description: Number of subjects to experience bleeding defined as Bleeding Academic Research Consortium (BARC) 1, 2, 3 or 5 or EASY hematoma classification after transradial/ulnar procedures (I-V)
Time Frame: From date of randomization until the date of first documented bleeding event up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target
Number analyzed (Participants) | 61 | 60 | 57
Participants | 14 | 15 | 15

2. Primary Outcome: Adverse Clinical Events
Description: Number of subjects to experience a Net Adverse Clinical Event (NACE) defined as all-cause mortality, myocardial infarction, stroke, target lesion revascularization, or major bleeding
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target
Number analyzed (Participants) | 61 | 60 | 57
Participants | 2 | 0 | 2

3. Secondary Outcome: Stent Thrombosis
Description: Number of subjects to experience stent thrombosis
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target
Number analyzed (Participants) | 61 | 60 | 57
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately one month on all participants.
Arm/Group | Low ACT Target | Medium ACT Target | High ACT Target
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 4/61 | 5/61 | 8/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low ACT Target (N=61) | Medium ACT Target (N=61) | High ACT Target (N=58)
Vessel Closure (Surgical and medical procedures) | 0 (0) | 1 (1) | 2 (2)
Dissection (Surgical and medical procedures) | 3 (3) | 4 (4) | 6 (6)
Spasm (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03772613/Prot_SAP_000.pdf